CLINICAL TRIAL: NCT04876742
Title: A Randomised Placebo-controlled Double-blind Exploratory Trial Within Cohort Using Wheat Beer for Prevention of Delirium in Intensive Care Patients
Brief Title: Wheat Beer for Prevention of Delirium in Intensive Care Patients
Acronym: BABE-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BASEC 2022-00779
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: ICU Delirium
MeSH Terms: interventions — Beer; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.5 liters of alcoholic beer (Experimental)
  Interventions: Other: Beer
- 0.5 liters of water (Placebo Comparator)
  Interventions: Other: Water
- non-interventional cohort control group (No Intervention)

INTERVENTIONS:
Other: Beer — As interventive agent 0.5 L organic alcohol-containing wheat beer produced by the brewery "Unser Bier" in Basel, Switzerland, is administered once a day at 8pm for 6 consecutive days after enrolment.
  Arms: 0.5 liters of alcoholic beer
Other: Water — For the interventional control group 0.5L water is administered once a day at 8pm for 6 consecutive days after enrolment.
  Arms: 0.5 liters of water

SUMMARY:
The investigators hypothesise that the daily administration of 0.5L alcohol-containing wheat beer at 8 pm over a study period of 6 days in a row leads to a lower prevalence of delirium compared to water following the same administration scheme.

DETAILED DESCRIPTION:
Delirium

Delirium is a complex state of confusion that can be seen as an acute failure of brain function. It is characterised by fluctuating deficits in cognition and attention, dysregulation of emotions and circadian rhythm as well as psychomotor changes.

In intensive care units (ICU) delirium is the most frequent syndromic complication with a prevalence between 26 - 60%. In mechanically ventilated patients, delirium is even detected in more than 80%. In elective cardiac surgery patients admitted to the ICU for postoperative monitoring postoperative delirium presents as a major complication and occurs in up to 33.5%. Hypoactive delirium outperforms the other two types - hyperactive and mixed - by far.

Occurrence of delirium is associated with several negative repercussions: Delirious patients show higher prevalence in morbidity and mortality, longer stays in intensive care units and the regular ward, as well as impaired cognitive function even months after the acute illness. The intensity of impairment in cognitive and executive function correlates with the duration of delirium. Furthermore, delirious patients cause major additional costs of up to 20% more compared to non-delirious patients.

Although there are several approaches for prevention of deliria in ICUs they are still highly prevalent causing a high and versatile burden as mentioned above. The several mainly pharmacological treatment approaches are more to be seen as a symptomatic treatment than a causal treatment. No groundbreaking prevention or treatment strategy has been found so far. Therefore, improvement of existing and development of new prevention strategies is therefore crucial and highly necessary. Further it has to be shown if prevention of delirium has an effect on clinical outcome.

Between March 2018 and February 2019, 584 patients that met the inclusion criteria of this study were admitted to the ICU of the University Hospital Basel. Of those, 167 patients (28.6%) developed a delirium within the first 48 hours. After 7 days (168 hours), 277 (47%) had at least once an ICDSC score of ≥4.

Wheat beer

Consumption of alcoholic beverages and therewith beer is widespread in Switzerland. Healthy effects of moderate beer consumption, especially benefits for prevention of cardiovascular diseases, are discussed in literature. Beer's major ingredients are water, hop, malt and yeast.

Alcohol Surveys in US American ICUs showed a pre-existing alcohol use disorder in 16-31% of ICU patients. Further research showed anamnestic alcohol abuse as a significant risk factor for development of delirium in ICUs.

Swiss governmental statistics show a widespread alcohol consumption among the Swiss population: While 82% consume alcohol periodically, 10% drink alcoholic beverages on a daily and almost 60% at least on a weekly basis. Alcohol consumption increases with age. In the group of the over 75-year-olds around 40% drink alcohol daily. Around 5% of the population bear a chronic risky alcohol consumption, 16% get drunk at least once a month. Thereby beer is one of the most popular beverages.

Alcohol, in alcoholic beverages ethanol, targets multiple central receptors and neural networks. In habituated individuals an abrupt abstinence from alcohol consumption leads to generalised central hyperexcitability due to unchecked excitation and impaired inhibition whereby alcohol withdrawal syndrome (AWS) and delirium tremens (DT) are more likely to occur. Similar mechanisms can be thought of in patients with moderate, non-abusive alcohol consumption favouring or causing delirium.

Hop Hop (Humulus lupulus) is a major ingredient of beer. Its main pharmacologically active constituent is humulone. It bears several health beneficial properties. Its main impact is the calming effect, which could be shown in a study in healthy nurses when consuming alcohol-free beer. Improvement of sleep quality and a hypnagogic effect induced by alcohol-free beer and hop extracts could also be shown in different studies.

On the molecular level the hop's sedating and hypnotic effect could be shown at the gamma-aminobutyric acid A (GABAA) receptor in a rat model which - positively modulated by ethanol - shortened sleep onset, increased duration of sleep and decreased the spontaneous locomotion.

Standard procedure and treatment of delirium at University Hospital Basel (USB)

All patients admitted to the ICU receive a standard care prevention for delirium including management of causes of delirium such as pain treatment using non-opioid and opioid analgesics and support of sleep-wake-cycle using Melatonin (Circadin®). The support in perception, orientation and communication as well as early and regular mobilisation, general stress reduction and inclusion of patient's next of kin are the main pillars of standard delirium care prevention.

For assessment of delirium Richmond Agitation Sedation Scale (RASS) and the Intensive Care Delirium Screening Checklist (ICDSC) are used regularly for delirium recognition (see "Measurement of delirium and sedation" in section 3.2 for details).

Current standard prevention and treatment of non-withdrawal delirium in the intensive care unit of the University Hospital Basel depends on the type of delirium.

Hyperactive and mixed delirium (ICDSC ≥ 4, RASS > 0) is treated when RASS ≥ 2 with Quetiapin (Seroquel®) orally or Haloperidol (Haldol®) intravenously if oral administration is not possible. As rescue for excessive motoric restlessness Levomepromazin-neuraxpharm intravenous or intramuscular is used. If restlessness with RASS ≥ 2 is persistent, syringe pumps with Dexmedetomidine (Dexdor®) or Propofol (Propofol®) are installed.

For treatment of hypoactive delirium, caring measures including registering and rapid handling of hunger, thirst, urine or stool urging are of great importance. Further preventive measures of delirium in general are applied for treatment such as giving orientation and feeling of safety, support of perception, activation and mobilisation.

For withdrawal delirium a separate treatment algorithm is provided. According to the intern treatment concept withdrawal delirium presents usually as hyperactive delirium with agitation tremor, tachycardia, sweating and hallucination in combination. For the prevention and treatment the same non-pharmacological procedures as described above for other types of deliria are applied.

Pharmacologically Lorazepam (Temesta®) or Phenobarbital is administered in case of motoric agitation. In case of conducting oneself in an endangering way for the patient itself or others a Propofol perfusor might be installed. Additionally, Clonidine (Catapressan®) is administered when strong vegetative symptoms occur. As a rescue treatment for most intense motoric agitation Levomepromazin-neuraxpharm is administered. For concomitant psychosis Haloperidol (Haldol®) is foreseen for its treatment. Alongside an early start of nutritional therapy as well as substitution of vitamins and minerals are important.

Research question

The BABE-D clinical trial wants to provide answers to the question if delirium in critically ill patients can be prevented or reduced in duration, as well as if intensity of agitation can be reduced by regularly administering a moderate amount of beer.

ELIGIBILITY:
Inclusion criteria

All Patients meeting the following criteria are eligible for the study:

* Risk of delirium: ICU patients with expected length of stay (LOS) ≥ 24 hours
* Naso-gastric tube in situ
* ICU stay ≤ 72h until first study intervention
* Women: negative pregnancy test, age ≥50 years or status post hysterectomy/bilateral ovariectomy
* Adult patients (age ≥ 18 years)
* ≥ 50 kg body weight or BMI ≥18.5

Exclusion Criteria

Patients fulfilling the following criteria are excluded from the study:

* Pre-existing liver pathologies
* Patients after bone marrow transplantation
* Women: breastfeeding
* Pre-existing delirium (ICDSC ≥ 4)
* Terminal state
* Active psychosis
* Anamnestic complete alcohol abstinence or status post alcohol abuse
* Especially vulnerable patients
* Allergy to any ingredient(s) of beer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of delirium | 7 days
  Development of delirium until day 7 after enrolment

SECONDARY OUTCOMES:
Delirium-free days | 30 days
  Delirium-free days alive
Sedation-free days | 30 days
  Sedation-free days alive
Agitation-free days | 30 days
  Agitation-free days alive

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the data through a controlled access repository. The data sharing plan may be provided. In addition, anonymised data will be shared upon request.
Supporting Information: Study Protocol, ICF
Time Frame: As soon as legally and ethically possible after trial publication.
Access Criteria: Anyone interested can contact the study team and wherever legally and ethically possible data will be shared. Additional supporting information may as well be shared upon request.